CLINICAL TRIAL: NCT06127212
Title: Bioequivalence Study of Dapagliflozin 10 mg Film-coated Tablet Produced by PT Dexa Medica in Comparison With the Comparator Drug (Forxiga® 10 mg Film-Coated Tablet, Manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China Imported by PT AstraZeneca Indonesia, Indonesia)
Brief Title: Bioequivalence Study of Dapagliflozin 10 mg Film-coated Tablets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: PT Equilab International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE. 754/EQL/2022
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This was a bioequivalence study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Dapagliflozin Dexa Medica (Experimental): Dapagliflozon 10 mg Film-Coated tablet, produced by PT Dexa Medica, Indonesia.
  Interventions: Drug: Dapagliflozin 10 mg film-coated tablet
- Reference Forxiga AstraZeneca (Active Comparator): Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia.
  Interventions: Drug: Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia

INTERVENTIONS:
Drug: Dapagliflozin 10 mg film-coated tablet — One tablet of the test drug was given orally (swallowed with 240 mL of 20% glucose solution in water), after an overnight fast.
  Other Names: Test
  Arms: Test Dapagliflozin Dexa Medica
Drug: Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia — One tablet of the reference drug was given orally (swallowed with 240 mL of 20% glucose solution in water), after an overnight fast.
  Other Names: Reference
  Arms: Reference Forxiga AstraZeneca

SUMMARY:
The study was an open-label, randomized, single-dose, two-period, two-sequence, two-day crossover study, conducted to find out whether the dapagliflozin 10 mg film-coated tablet produced by PT Dexa Medica (test drug) was bioequivalent to the reference drug (Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia), under fasting condition with a five days wash-out period, involving 24 healthy adult male and female subjects.

DETAILED DESCRIPTION:
The study was an open-label, randomized, single-dose, two-period, two-sequence, two-day crossover study, conducted to find out whether the dapagliflozin 10 mg film-coated tablet produced by PT Dexa Medica (test drug) was bioequivalent to the reference drug (Forxiga® 10 mg Film-Coated Tablet, manufactured by AstraZeneca Pharmaceuticals LP, USA for AstraZeneca Pharmaceuticals Co. Ltd., China imported by PT AstraZeneca Indonesia, Indonesia), under fasting condition with a five days wash-out period, involving 24 healthy adult male and female subjects. The participating subjects had an overnight fast and in the next morning were given orally either one film-coated tablet of the test drug or one film-coated tablet of the reference drug with a total 240 mL of a 20% glucose solution in water. Following drug administration, 60 mL of 20% glucose solution was administered at every 15 minutes for up to 4 hours after dosing as maintenance to prevent hypoglycemic symptoms. Blood samples were drawn before taking the drug (control) and at 0.25, 0.50, 0.75, 1.00, 1.25, 1.50,1.75, 2.00, 3.00, 4.00, 6.00, 8.00, 12.00, 24.00, 36.00 and 48.00 hours after drug administration. The blood samples were analyzed to investigate the pharmacokinetics parameters of the single dose administration of dapagliflozin. The plasma concentrations of dapagliflozin were determined by using a validated ultra-performance liquid chromatography with tandem mass spectroscopy detection (UPLC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
2. Healthy male and female subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening and could be considered healthy based on the evaluation.
3. Aged 18 - 55 years inclusive.
4. Preferably non-smokers or smoke less than 10 cigarettes per day.
5. Body mass index within 18 to 25 kg/m2
6. Vital signs (after 10 minutes rest) must be within the following ranges:

   * Systolic blood pressure: 100 - 129 mmHg
   * Diastolic blood pressure: 60 - 84 mmHg
   * Pulse rate: 60 - 90 bpm.
7. Willing to practice abstention or contraception during the study

Exclusion Criteria:

1. History of allergy or hypersensitivity or contraindication to dapagliflozin or allied drugs.
2. Pregnant or lactating female (urinary pregnancy test was applied to female subjects at screening and before taking the study drug).
3. Any major illness in the past 90 days or clinically significant ongoing chronic medical illness.
4. Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver function test (AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin ≥ 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL and ureum ≥ 1.5 ULN), etc.
5. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
6. Positive result for COVID-19 rapid antigen test.
7. Clinically significant hematology abnormalities.
8. Clinically significant electrocardiogram (ECG) abnormalities.
9. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery.
10. Past history of anaphylaxis or angioedema.
11. History of drug or alcohol abuse within 12 months prior to screening for this study.
12. Participation in any clinical trial within the past 90 days calculated from the last visit until this study's first dosing day.
13. History of any bleeding or coagulative disorders.
14. Presence of difficulty in accessibility of veins in left or right arm.
15. A donation or significant blood loss within 90 days before this study's first dosing day.
16. Intake of any prescription (especially dapagliflozin and empagliflozin), non-prescription drug (including hormonal contraception), food supplements or herbal medicines within 21 days of this study's first dosing day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | 48 hours
  Area under the plasma concentration-time curve to the last observer quantifiable concentration at time t
Cmax | 48 hours
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUC(0-inf) | 48 hours
  Area under the plasma concentration-time curve extrapolated to infinitive time
T1/2 | 48 hours
  Plasma half-life
Tmax | 48 hours
  Time taken to reach maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Danang A Yunaidi, MD, Principal Investigator — Equilab International
Locations (1):
- PT Equilab International, Jakarta, Indonesia